CLINICAL TRIAL: NCT06567834
Title: Clinical Evaluation of Violet Light Filtration and High-resolution Lathing on a Diffractive Extended Depth of Focus Intraocular Lens (IOL)
Brief Title: Clinical Evaluation and Comparison of the Tecnis Symfony Optiblue and Tecnis Symfony IOLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Empire Eye and Laser Center (Other)
Collaborators: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Daniel H. Chang, MD, Principal Investigator, Empire Eye and Laser Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMP-2022-001
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Cataract; Presbyopia
Keywords: Extended Depth of Focus IOLs; Dysphotopsia; Low Contrast Vision; Presbyopia Correction; Halos; Starbursts
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomly assigned 1:1 to bilateral implantation with either Tecnis Symfony Optiblue/Tecnis Symfony Optiblue Toric (ZXR00V/ZXW150) or Tecnis Symfony/Tecnis Symfony Toric (ZXR00/ZXT150).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tecnis Symfony Optiblue (Experimental): Tecnis Symfony Optiblue/Tecnis Symfony Optiblue Toric (ZXR00V/ZXW150)
  Interventions: Device: Tecnis Symfony Optiblue/Tecnis Symfony Optiblue Toric (Models ZXR00V/ZXW150)
- Tecnis Symfony (Active Comparator): Tecnis Symfony/Tecnis Symfony Toric (ZXR00/ZXT150)
  Interventions: Device: Tecnis Symfony/Tecnis Symfony Toric (Models ZXR00/ZXT150)

INTERVENTIONS:
Device: Tecnis Symfony Optiblue/Tecnis Symfony Optiblue Toric (Models ZXR00V/ZXW150) — Multifocal IOL with violet light filtration and high-resolution lathing
  Arms: Tecnis Symfony Optiblue
Device: Tecnis Symfony/Tecnis Symfony Toric (Models ZXR00/ZXT150) — Multifocal IOL with ultraviolet filtration
  Arms: Tecnis Symfony

SUMMARY:
The goal of this clinical study is to compare the Tecnis Symfony Optiblue intraocular lens implant to the Tecnis Symfony intraocular lens implant in patients over 22 years old with cataracts in both eyes. The main questions it aims to answer are:

Which lens has less nighttime side effects? Which lens has higher patient satisfaction?

Participants will undergo a minimum of 7 study visits where they will complete a variety of vision tests and vision questionnaires.

DETAILED DESCRIPTION:
This is 6 month, prospective, single center, subject/evaluator masked, bilateral, randomized clinical investigation of the TECNIS Symfony Model ZXR00V/ ZXW150 IOLs versus the TECNIS Symfony Model ZXR00/ZXT150 control IOL.

The study will enroll approximately 60 subjects to achieve approximately 54 randomized and bilaterally implanted subjects, resulting in approximately 25 evaluable subjects in each lens group at 6 months. Subjects are to be implanted with the same IOL in both eyes, the ZXR00V/ZXW150 or the ZXR00/ ZXT150 control IOL. The eye implanted first will be considered the primary study eye.

Surgeons will perform routine, small-incision cataract surgery and implant the study lenses using an implantation system qualified by the respective manufacturer for use with that IOL. The target for refractive outcomes will be emmetropia for both eyes.

All subjects will undergo a minimum of 7 study visits: Preoperative for both eyes; Operative for each eye; 1 week first eye and second eye, 1 month and 6 month visits for both eyes together.

The primary endpoint is patient reported nighttime dysphotopsia symptoms as measured by the PRVSQ v2 questionnaire.

The secondary endpoints are 25% low contrast visual acuity with glare and patient satisfaction.

OTHER ENDPOINTS

* Monocular photopic uncorrected distance visual acuity (UCDVA)
* Binocular UCDVA and uncorrected near visual acuity (UCNVA) at 40 cm
* 10% and 25% low contrast acuity without glare
* Residual refractive error
* Natural binocular reading distance
* Distance of subjective near blur
* Lens findings/complications
* Spectacle use
* Other ocular/visual symptoms (non-directed chief complaint)
* Patient satisfaction and recommendation
* Time with physician in exam room

ELIGIBILITY:
Inclusion Criteria:

* All criteria apply to each study eye

  * Minimum 22 years of age
  * Bilateral cataracts for which posterior chamber IOL implantation has been planned
  * Preoperative best corrected distance visual acuity (BCDVA) of 20/40 Snellen or worse with a glare source or 20/40 Snellen or worse without a glare source
  * Potential for postoperative BCDVA of 20/30 Snellen or better
  * Corneal astigmatism:
  * Normal corneal topography
  * Preoperative corneal astigmatism range from 0 D - 2.0 D
  * Clear intraocular media other than cataract in each eye
  * Availability, willingness, and sufficient cognitive awareness to comply with examination procedures
  * Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries
  * Ability to understand and respond to a questionnaire in English

Exclusion Criteria:

* All criteria apply to each study eye:

  * Requiring an intraocular lens power outside the available range of power
  * Any clinically significant pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils)
  * Irregular corneal astigmatism
  * Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
  * Prior corneal refractive surgery (LASIK, LASEK, radial keratotomy (RK), photorefractive keratectomy (PRK), etc.) or intraocular surgery. Note: Prophylactic peripheral iridotomies and peripheral laser retinal repairs that, in the opinion of the investigator will not confound study outcomes or increase risk to the subject, are acceptable.
  * Corneal abnormalities such as stromal, epithelial, or endothelial dystrophies that are predicted to cause visual acuity losses to a level worse than 20/30 Snellen during the study
  * Inability to achieve keratometric stability for contact lens wearers
  * Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
  * Subject with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
  * Use of systemic or ocular medications that may affect vision
  * Prior, current, or anticipated use during the course of the 6 month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
  * Poorly controlled diabetes
  * Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.). Note: controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable.
  * Known ocular disease or pathology that, in the opinion of the investigator,
  * may affect visual acuity
  * may require surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, uncontrolled glaucoma, etc.)
  * may be expected to require retinal laser treatment or other surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
  * Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
  * Concurrent participation or participation within 60 days prior to preoperative visit in any other clinical trial
  * Desire for monovision correction

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Patient reported nighttime dysphotopsia symptoms | Pre-op visit, 1 month post-op visit, 6 month post-op visit
  Patient-Reported Visual Symptoms Questionnaire (PRVSQ)

SECONDARY OUTCOMES:
Low contrast visual acuity with glare | 1 month post-op visit, 6 month post-op visit
  Mesopic 25% low contrast visual acuity with glare
Patient overall satisfaction | 1 month post-op visit, 6 month post-op visit
  Patient Recommendation Questionnaire

OTHER OUTCOMES:
Monocular photopic UCDVA | Pre-op visit
  Uncorrected distance visual acuity (UCDVA) - photopic, monocular (Snellen visual acuity)
Monocular photopic UCDVA | 1 week post-op visit first and second eye, 1 month post-op visit, 6 month post-op visit
  Uncorrected distance visual acuity (UCDVA) - photopic, monocular (The Early Treatment Diabetes Retinopathy Study (ETDRS) visual acuity) ETDRS letters range from 58.18 mm to 2.92 mm in height, corresponding to Snellen visual acuity fractions of 20/200 to 20/10, respectively. The larger the number, the worse the visual acuity.
Binocular UCDVA | 1 month post-op visit, 6 month post-op visit
  Uncorrected distance visual acuity (UCDVA) - photopic, binocular (The Early Treatment Diabetes Retinopathy Study (ETDRS) visual acuity) ETDRS letters range from 58.18 mm to 2.92 mm in height, corresponding to Snellen visual acuity fractions of 20/200 to 20/10, respectively. The larger the number, the worse the visual acuity.
UCNVA at 40 cm | 1 month post-op visit, 6 month post-op visit
  Uncorrected near visual acuity (UCNVA) - photopic, binocular at 40 cm (The Early Treatment Diabetes Retinopathy Study (ETDRS) visual acuity) ETDRS letters range from 58.18 mm to 2.92 mm in height, corresponding to Snellen visual acuity fractions of 20/200 to 20/10, respectively. The larger the number, the worse the visual acuity.
Low contrast acuity without glare | 1 month post-op visit, 6 month post-op visit
  10% and 25% low contrast acuity without glare (photopic and mesopic)
Residual refractive error | 1 week post-op visit first and second eye, 1 month post-op visit, 6 month post-op visit
  Best corrected distance visual acuity (BCDVA) - photopic, monocular
Natural binocular reading distance | 1 month post-op visit, 6 month post-op visit
  Natural binocular reading distance (cm)
Distance of subjective near blur | 1 month post-op visit, 6 month post-op visit
  Distance of subjective near blur (cm)
Lens findings/complications | 1 day post-op visit first and second eye, 1 week post-op visit first and second eye, 1 month post-op visit, 6 month post-op visit
  Biomicroscopic slit-lamp exam including determination of medical and lens findings/complications
Spectacle use | 1 month post-op visit, 6 month post-op visit
  Patient-Reported Spectacle Independence Questionnaire (PRSIQ)
Other ocular/visual symptoms (non-directed chief complaint) | 1 week post-op visit first and second eye, 1 month post-op visit, 6 month post-op visit
  A comprehensive list of all other self-reported ocular/visual complaints, in the patient's own words, will be compiled
Patient satisfaction and recommendation | 1 month post-op visit, 6 month post-op visit
  Patient Recommendation Questionnaire
Time with physician in exam room | 1 day post-op visit first and second eye, 1 week post-op visit first and second eye, 1 month post-op visit, 6 month post-op visit
  Time with physician in exam room (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Chang, MD, Principal Investigator — Empire Eye and Laser Center
Locations (1):
- Empire Eye and Laser Center, Bakersfield, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang DH, Janakiraman DP, Smith PJ, Buteyn A, Domingo J, Jones JJ, Christie WC. Visual outcomes and safety of an extended depth-of-focus intraocular lens: results of a pivotal clinical trial. J Cataract Refract Surg. 2022 Mar 1;48(3):288-297. doi: 10.1097/j.jcrs.0000000000000747. PMID 34269326
- [Background] Hammond BR, Sreenivasan V, Suryakumar R. The Effects of Blue Light-Filtering Intraocular Lenses on the Protection and Function of the Visual System. Clin Ophthalmol. 2019 Dec 5;13:2427-2438. doi: 10.2147/OPTH.S213280. eCollection 2019. PMID 31824137
- [Background] Chang DH, Pastuck T, Rosen R, Hollmann S, Babic T, Stapars A. Violet and Blue Light: Impact of High-Energy Light on Vision and Health. (2020) Violet and Blue Light: Impact of High-Energy Light on Vision and Health. J Ophthalmic Stud 3(2):1-8. dx.doi.org/10.16966/2639-152X.119
- [Background] Chang DH, Thompson VM, Christie WC, Chu YR, Vida RS. Clinical Evaluation of a Modified Light Transmission Short-Wavelength Filtering Intraocular Lens Compared to a Colorless Control. Ophthalmol Ther. 2023 Jun;12(3):1775-1785. doi: 10.1007/s40123-023-00709-w. Epub 2023 Apr 18. PMID 37071325
- [Background] Zhang L, Lin D, Wang Y, Chen W, Xiao W, Xiang Y, Zhu Y, Chen C, Dong X, Liu Y, Chen W, Lin H. Comparison of Visual Neuroadaptations After Multifocal and Monofocal Intraocular Lens Implantation. Front Neurosci. 2021 Jun 14;15:648863. doi: 10.3389/fnins.2021.648863. eCollection 2021. PMID 34194292
- [Background] van der Mooren M, Alarcon A, Jenkins Sanchez MD, Chang DH. Effect of Violet Light-Filtering and Manufacturing Improvements in an Extended Depth-of-Focus Intraocular Lens on Visual Performance. Clin Ophthalmol. 2023 Mar 1;17:701-709. doi: 10.2147/OPTH.S396823. eCollection 2023. PMID 36891506
- [Background] Chang DH, Waring GO, Hom M, Barnett M. Presbyopia Treatments by Mechanism of Action: A New Classification System Based on a Review of the Literature. Clin Ophthalmol. 2021 Sep 6;15:3733-3745. doi: 10.2147/OPTH.S318065. eCollection 2021. PMID 34522079
- [Background] Chang DH, Hu JG, Lehmann RP, Thompson VM, Tsai LH, Thomas EK. Clinical performance of a hybrid presbyopia-correcting intraocular lens in patients undergoing cataract surgery in a multicenter trial. J Cataract Refract Surg. 2023 Aug 1;49(8):840-847. doi: 10.1097/j.jcrs.0000000000001205. PMID 37097283
- [Background] de Silva SR, Evans JR, Kirthi V, Ziaei M, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2016 Dec 12;12(12):CD003169. doi: 10.1002/14651858.CD003169.pub4. PMID 27943250
- [Background] Han KE, Lee JE. Comparative Evaluation of Visual Performance and Patient Satisfaction following Cataract Surgery: A Retrospective Analysis of an Extended Depth-of-Focus Intraocular Lens and a Diffractive Multifocal Lens with Extended Depth of Focus. J Clin Med. 2023 Nov 28;12(23):7368. doi: 10.3390/jcm12237368. PMID 38068421
- [Background] Woodward MA, Randleman JB, Stulting RD. Dissatisfaction after multifocal intraocular lens implantation. J Cataract Refract Surg. 2009 Jun;35(6):992-7. doi: 10.1016/j.jcrs.2009.01.031. PMID 19465282
- [Background] Ntonti P, Bakirtzis M, Delibasis K, Seimenis I, Tsinopoulos I, Labiris G. Impact of personality on the decision process and on satisfaction rates in pseudophakic presbyopic correction. J Cataract Refract Surg. 2022 Dec 1;48(12):1433-1439. doi: 10.1097/j.jcrs.0000000000001021. PMID 35862830
- [Background] Kim EC, Cho SY, Kang JE, Nam G, Yoon YC, Whang WJ, Na KS, Kim HS, Hwang HS. Comparative Analysis of Optical Quality of Monofocal, Enhanced Monofocal, Multifocal, and Extended Depth of Focus Intraocular Lenses: A Mobile Model Eye Study. Transl Vis Sci Technol. 2023 Jul 3;12(7):5. doi: 10.1167/tvst.12.7.5. PMID 37405796
- [Background] Meikies D, van der Mooren M, Terwee T, Guthoff RF, Stachs O. Rostock Glare Perimeter: a distinctive method for quantification of glare. Optom Vis Sci. 2013 Oct;90(10):1143-8. doi: 10.1097/OPX.0b013e318295a720. PMID 23811606
- [Background] Hays RD, MacRae S, Holladay J, Tarver ME, Lum F, Stark W, Weidmer B, Kumar N, Lau G, Nguyen T, Schallhorn S, Eydelman M, Masket S. Development of a Patient-Reported Outcome Measure to Assess Symptoms Associated with Cataract Surgery and Intraocular Lens Implants. Ophthalmology. 2023 Jul;130(7):715-725. doi: 10.1016/j.ophtha.2023.02.026. Epub 2023 Apr 12. PMID 37055289
- [Background] Masket S, Lum F, MacRae S, Hays RD, Tarver ME, Holladay J, Yoon G, Nguyen T, Stark W, Kumar N, Lau G, Schallhorn S, Eydelman M. Symptoms and Satisfaction Levels Associated with Intraocular Lens Implants in the Monofocal and Premium IOL Patient-Reported Outcome Measure Study. Ophthalmology. 2023 Jul;130(7):726-734. doi: 10.1016/j.ophtha.2023.02.027. Epub 2023 Apr 15. PMID 37061911
- [Background] Aslam TM, Dhillon B, Tallentire VR, Patton N, Aspinal P. Development of a forced choice photographic questionnaire for photic phenomena and its testing - repeatability, reliability and validity. Ophthalmologica. 2004 Nov-Dec;218(6):402-10. doi: 10.1159/000080944. PMID 15564759
- [Derived] Chang DH, Kao AA, Huggins LK, Albert JN, Whinery JN, Camirand BM. Clinical Evaluation of Violet Light Filtration and High-Resolution Lathing on a Diffractive Extended Depth of Focus IOL. Ophthalmol Ther. 2024 Dec;13(12):3135-3147. doi: 10.1007/s40123-024-01056-0. Epub 2024 Oct 25. PMID 39455493